CLINICAL TRIAL: NCT02025374
Title: The Comparison of Hyperbaric Bupivacaine Plus Fentanyl and Hyperbaric Levobupivacaine Plus Fentanyl Administered Intrathecally in Patients Undergoing Elective Cesarean Section
Brief Title: Hyperbaric Bupivacaine and Hyperbaric Levobupivacaine in C/S
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Ozlem Sagir, MD, Assistant Professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: osagir1
Record Dates: First submitted 2013-12-12; First posted 2014-01-01 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Health Care; Drugs
Keywords: spinal anesthesia; cesarean section; hyperbaric levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperbaric levobupivacaine (Experimental): Group 2 Hyperbaric levobupivacaine % 0.5 plus fentanyl; 2 ml total intrathecally
  Interventions: Drug: Hyperbaric levobupivacaine
- Hyperbaric bupivacaine (Active Comparator): Group 1 Hyperbaric bupivacaine % 0.5 plus fentanyl 2 ml intrathecally
  Interventions: Drug: Hyperbaric bupivacaine % 0.5

INTERVENTIONS:
Drug: Hyperbaric levobupivacaine
  Other Names: Chirocaine %0.75
  Arms: Hyperbaric levobupivacaine
Drug: Hyperbaric bupivacaine % 0.5
  Other Names: Marcaine heavy % 0.5
  Arms: Hyperbaric bupivacaine

SUMMARY:
Aim of the Study To compare the effects of hyperbaric bupivacaine plus fentanyl with hyperbaric levobupivacaine plus fentanyl on spinal block quality, haemodynamics and need for analgesics in patients undergoing elective cesarean section. Our hypothesis is that hyperbaric levobupivacaine will provide equal block quality, but better haemodynamic conditions compared to hyperbaric bupivacaine.

DETAILED DESCRIPTION:
Material - Method 60 patients, American Society of Anesthesiology (ASA) group I-II, between the ages of 18-45 who were scheduled for elective cesarian section under regional anesthesia are going to be included. Patients with contraindications to regional anesthesia, known allergy, suffering from pregnancy induced hypertension or placenta previa will be excluded from the study.

Patients will not be premedicated. After routine monitorization , IV access and fluid replacement patients will be separated to two groups on a randomised manner. Under sterile conditions spinal anesthesia will be performed in the sitting position at the level L3-4 or L 4-5 via epidural-spinal combined including a 27 G spinal needle.

Group 1 will receive 8 mg hyperbaric bupivacaine plus 20 mcg fentanyl /2ml intrathecally.

Group 2 will receive 8 mg hyperbaric levobupivacaine plus 20 mcg fentanyl/2ml intrathecally.

The Hyperbaric form of Levobupivacaine is not available on market , so it will be prepared with the addition of % 30 dextrose by another anesthesiologist who will be blinded to the patients.

Preparation: 2 ml of %0,75 levobupivacaine + 0,8 mL %30 dextrose + 0,2 mL of saline will be mixed. So it will contain 5 mg levobupivacaine and %8 dextrose per ml.

Hypotension will be defined as a decrease in blood pressure more than % 30 percent of the basal measured systolic arterial pressure. Hypotension will be treated with 250 ml fast saline infusion and if no response with 5 mg of ephedrine IV. A heart rate under 50 beats/min will be defined as bradycardia and will be treated with 0.5 mg atropine i.v.. If the anesthesia is not sufficient 10 ml of % 0.25 levobupivacaine wil be administered through the epidural catheter. The level of sensory and motor block will be evaluated and recorded every 3 minutes at the beginning and after 15 minutes it will be checked every 5 minutes until the end of surgery. Maximum level of sensory block, time to reach T4 dermatome and time to regression of 2 segments will be recorded. Nausea-vomiting, pruritus and shivering will also be recorded. Baby delivery time, which will be defined as the time from spinal medication to clamping of the umbilical cord will also be recorded. Total time of surgery will also be recorded. The time for the first analgesic requirement will be noticed as well. Patient and surgeon satisfaction will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

elective cesarean section no other coexisting medical situation

Exclusion Criteria:

known contraindication to regional anesthesia coexisting pregnancy induced problem placental mislocation known allergy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
evaluation of the changes in mean arterial blood pressure between two groups. | 6 month

SECONDARY OUTCOMES:
Time to reach T4 dermatome | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Balıkesir University Faculty of Medicine, Balıkesir, Turkey (Türkiye)